CLINICAL TRIAL: NCT04279912
Title: A Feasibility and Safety Clinical Trial of the Magnetic Resonance Guided Focused Ultrasound (MRgFUS) for the Management of Tremor in Patients With Multiple Sclerosis
Brief Title: MR-Guided Focused Ultrasound (MRgFUS) for the Management of Tremor in Patients With Multiple Sclerosis
Acronym: MSFUS001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Neurosurgeon, Principal Investigator, Assistant Professor, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 029-2019
Record Dates: First submitted 2020-01-31; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Tremor; Multiple Sclerosis; MR-guided Focused Ultrasound
MeSH Terms: conditions — Multiple Sclerosis; Tremor

STUDY DESIGN:
Intervention Model Description: Single-centre, prospective, single-arm, open-label pilot trial assessing the feasibility and safety of MRgFUS thalamotomy for refractory hand tremor in up to 6 patients with multiple sclerosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Multiple Sclerosis and Tremor (Experimental): Participants will undergo MRgFUS thermal ablation of the ventral intermedius (Vim) thalamus contralateral to the most affected side of the body.
  Interventions: Device: Focused Ultrasound (MRgFUS) for the Management of Tremor in Patients With Multiple Sclerosis

INTERVENTIONS:
Device: Focused Ultrasound (MRgFUS) for the Management of Tremor in Patients With Multiple Sclerosis — The intervention is MRIgFUS thermal ablation of the ventral intermedius (Vim) thalamus contralateral to the most affected side of the body.

SUMMARY:
This study will be a single-centre, prospective, single-arm, open-label pilot trial assessing the feasibility and safety of unilateral MR-guided focused ultrasound (MRgFUS) thalamotomy for refractory hand tremor in up to 12 patients with multiple sclerosis (relapsing-remitting, primary progressive or secondary progressive MS). This study will be conducted at the Focused Ultrasound Centre of Excellence and MS Clinic located at Sunnybrook Health Sciences Centre/ University of Toronto. Patients with stable MS and refractory hand tremor providing informed consent will receive MRgFUS thermal ablation of the Vim thalamus contralateral to the most affected side of the body (frequently this will be the dominant hand).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18-80 years
* Willing and able to give consent and attend all study visits
* A confirmed diagnosis of medication-refractory, MS-related hand tremor
* No clinical evidence of relapse over 12 months or more before enrollment
* No MRI activity over 3 months or more before enrollment
* Presence of disabling postural or kinetic tremor
* Unsatisfactory tremor response to adequate trials of at least two medications
* Able to communicate sensations during the treatment
* Stable doses of all medications for 30 days prior to and during study

Exclusion Criteria:

* Severe cerebellar dysfunction measured by Scale for the Assessment and Rating of Ataxia (>35 out of 40)
* Severe weakness or sensory loss in arm contralateral to the side of the brain considered for MRgFUS
* Evidence of a superimposed or atypical movement disorder
* Unstable cardiac status such as angina pectoris, congestive heart failure, etc.
* Severe hypertension
* Patients with standard contraindications for MR imaging
* History of abnormal bleeding and/or coagulopathy
* Ischemic or hemorrhagic stroke within 6 months
* Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Untreated, uncontrolled sleep apnea
* Active or suspected acute or chronic uncontrolled infection
* Receiving anticoagulant or antiplatelet therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage within one month of MRgFUS surgery
* Not able or willing to tolerate the required prolonged stationary supine position during treatment
* Participating or have participated in another clinical trial in the last 30 days
* Unable to communicate with the investigator and staff
* Presence of neurodegenerative disease or significant cognitive impairment
* Presence of significant cognitive impairment (≤24 on MMSE)
* Uncontrolled major psychiatric disorder or suicidal ideation
* Risk factors for intraoperative or postoperative bleeding or documented coagulopathy
* Presence of brain tumours
* Any illness that in the investigator's opinion preclude participation in this study
* Pregnancy or lactation
* Legal incapacity or limited legal capacity
* Deep Brain Stimulation or a prior stereotactic ablation of the basal ganglia
* A history of seizures within the past year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Composite safety outcome of MRgFUS thalamotomy | 90 days
  Composite outcome of detectable Vim lesion on MRI scan; AND lack of new-onset or worsening of contralateral upper limb sensory loss or weakness

SECONDARY OUTCOMES:
Incidence and severity of adverse events related to MRgFUS thalamotomy | 1, 7, 30, 90 and 120 days
  Incidence and severity of adverse events possibly, probably or definitely related to the MRgFUS procedure at 1, 7, 30, 90 and 120 days after treatment.
Incidence and severity of adverse events related to MS disease relapse or progression | 30 and 90 days
  Incidence and severity of AEs possibly, probably or definitely-related to MS disease relapse or progression (based on clinical assessment) over 30 and 90 days.
Changes from baseline in the EDSS (Expanded Disability Status Scale) scores | 30 and 90 days
  Changes from baseline in the EDSS scores at 30 and 90 days. This is a scale to of quantify disability in multiple sclerosis. Score: 0 to 10 with higher scores meaning worse outcome.
Changes from baseline in the SARA (Scale for Assessment and Rating of Ataxia) scores | 30 and 90 days
  Changes from baseline in the SARA scores at 30 and 90 days. This is a scale to of quantify function and disability related to ataxia. Score: 0 to 40 with higher scores meaning worse outcome.
Changes from baseline in the speech intelligibility (percentage of intelligible words recorded during standardized passage reading) | 30 and 90 days
  Changes from baseline in intelligibility percentage at 30 and 90 days. Score: 0 to 100% with higher scores meaning better outcome.
Changes from baseline in QUEST (Quality of Life in Essential Tremor Questionnaire) scores | 30 and 90 days
  Changes from baseline in QUEST scores at 30 and 90 days. This is a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL) that generic QOL measures do not effectively capture, including activities of daily living that are affected by tremor. Higher scores mean worse outcome.
Change from baseline in the CRST (Clinical Rating Scale for Tremors) | 30 and 90 days
  Change from baseline in the treated upper limb tremor subscore of the CRST at 30 and 90 days. Score: 0 to 32 with higher scores meaning worse outcome.
Composite safety outcome of MRgFUS thalamotomy | 30 days
  Composite outcome of detectable Vim lesion on MRI scan; AND lack of new-onset or worsening of contralateral upper limb sensory loss or weakness

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Agessandro Abrahao, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No